CLINICAL TRIAL: NCT07237100
Title: A Pilot Study of Mirdametinib in Patients With Advanced Melanoma With an NF1 Mutation
Brief Title: Mirdametinib in Patients With Advanced NF1-mutant Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kevin Kim, MD (Other)
Responsible Party: Sponsor-Investigator, Kevin Kim, MD, Medical Director of Melanoma Clinical Research Program, Sutter Health
Organization: Sutter Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPMC24-MEL01
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Advanced Unresectable Melanoma; Metastatic Melanoma
Keywords: Neurofibromin 1 (NF1) mutation; advanced unresectable melanoma; Metastatic Melanoma; Melanoma; Mirdametinib
MeSH Terms: conditions — Melanoma; Neurofibromatoses | interventions — mirdametinib

STUDY DESIGN:
Intervention Model Description: The dosing schedule:
  • 4 mg BID for administered continuously (1 cycle = 28 days).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mirdametinib (Experimental): Patients receive mirdametinib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Mirdametinib

INTERVENTIONS:
Drug: Mirdametinib — Mirdametinib is a kinase inhibitor. It is taken by mouth twice a day
  Other Names: PD-0325901

SUMMARY:
The goal of this clinical trial is to evaluate clinical efficacy of mirdametinib in patients with advanced NF1-mutant melanoma whose disease has progressed while on or after previous immunotherapy. The main questions this study aims to answer are:

* To evaluate the feasibility of conducting a prospective single-center clinical trial of mirdametinib in patients with advanced NF1-mutant melanoma whose disease progresses during or after PD-1 antibody-based checkpoint inhibitor therapy.
* To evaluate preliminary clinical efficacy of mirdametinib in patients with advanced NF1-mutant melanoma whose disease has progressed while on or after previous immunotherapy
* To evaluate the safety profile of mirdametinib in patients with advanced NF1-mutant melanoma

DETAILED DESCRIPTION:
The purpose of this study is to test if mirdametinib is safe and effective in improving disease status and/or delaying progression of disease. Mirdametinib is being studied to see if it can help slow down or stop the growth of certain types of cancer.

Mirdametinib is a "MEK inhibitor," which targets specific pathways inside cancer cells. In some cancers, these pathways are overly active, causing the cells to grow and divide quickly. Mirdametinib is designed to block this activity, potentially slowing or stopping cancer growth.

Because mirdametinib is a targeted therapy, it focuses on the cancer cells more directly rather than attacking healthy cells throughout the body. This means it may work differently from traditional chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable or metastatic melanoma with an NF1 mutation; Variance of NF1 of unknown/ uncertain significance will not be eligible; The genetic analysis for somatic mutations must be performed in a lab that has obtained CLIA certification.
* Patients must have a report of NF1 sequencing analysis performed at CLIA-certified laboratory (by either tissue-based sequencing or liquid biopsy)
* Must have been previously treated with

  * anti PD-1/PD-L1 antibody; AND anti CTLA-4 antibody and/or anti LAG3 antibody;
  * UNLESS these standard checkpoint inhibitors are not clinically indicated or suitable (for example, comorbid conditions, such as autoimmune disease, or significant toxicity with prior checkpoint inhibitor treatment)
* Tumors must be progressing at the time of the enrollment
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Patients must be ≥ 18 years of age
* Patients must have measurable metastatic disease according to RECIST 1.1
* Patients must have adequate organ function, defined as follows:
* Absolute neutrophil count ≥ 1,500/μL
* Platelets ≥ 100,000/μL
* Hemoglobin ≥ 9 g/dL
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation. Estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m2 calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (Grade ≤1). • Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ 1 x ULN (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* Aspartate aminotransferase and alanine aminotransferase ≤ 3.0 x ULN (Grade ≤1) unless liver metastases are present, in which case they must be ≤ 5 x ULN (Grade ≤2).
* Adequate coagulation function, as determined by:
* International Normalized Ratio (INR) ≤ 1.5 × ULN (Grade ≤ 1). If the participant receives anticoagulant therapy, the INR > 1.5 × ULN is permitted, but the dose must be stable for at least 2 weeks before the start of the study treatments.
* PTT ≤ 1.5 × ULN.
* Adequate cardiac function, as determined by:
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg (Grade ≤ 2).
* LVEF ≥ 50% by MUGA or ECHO.
* No clinically significant ECG waveform abnormalities assessments at screening (one triplicate).
* Have normal serum calcium and phosphate levels (calcium level may be corrected for albumin level).
* Female patients are eligible to enroll and participate in the study if:
* Patient is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who:

  1. has had a hysterectomy.
  2. has had a bilateral oophorectomy (ovariectomy).
  3. has had bilateral tubal ligation.
  4. is postmenopausal (total cessation of menses for ≥1 year), OR
* Women of child-bearing potential must agree to use highly effective contraceptive methods (hormonal or barrier method of birth control or abstinence) during the trial period through at least six months after the last dose. Male patients or their partners must be surgically sterile or agree to use adequate contraception while receiving trial treatment and for three months thereafter. Contraceptive use by men or women should be consistent with Clinical Trials Coordination Group (CTCG) guidance.
* Patients must be able to understand the study procedures and agree to participate in the study by providing written informed consent.

Exclusion Criteria:

* Patients who were previously treated with MEK, ERK or RAF inhibitor therapy
* Patients with symptomatic brain metastasis or active brain lesions ≥ 6 mm size or those who require steroid treatment for brain lesions or leptomeningeal disease
* No systemic cancer therapy within 28 days of the study drug administration,
* Patients must not be simultaneously enrolled in any therapeutic clinical trial
* Patients must not have had investigational therapy administered ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing in this study.
* Patient has a history of, or evidence of, retinal pathology on ophthalmologic examination that is considered a risk factor for central serous retinopathy, retinal vein occlusion (RVO), or neovascular macular degeneration. Participants will be excluded from study participation if they have any of the following risk factors for RVO at Screening:

  * Intraocular pressure > 21 mmHg;
  * Serum cholesterol > 300 mg/dL;
  * Serum triglycerides > 300 mg/dL;
  * Hyperglycemia (fasting blood glucose > 125 mg/dL or random blood glucose > 200 mg/dL);
* History or current evidence of glaucoma or clinically significant abnormalities on the ophthalmological exam, including but not limited to cataract limiting the ability to examine the retina or any optical coherence tomography (OCT) finding that could be a significant risk factor for RVO, retinopathy or neovascular macular degeneration.

  o Note: Mild and controlled/stable age-related macular degeneration or non-proliferative diabetic retinopathy may be acceptable at the investigator's discretion after consultation with the ophthalmologist.
* History (within 6 months before the start of the study treatments) of clinically significant cardiac disease (New York Heart Association Class III or IV), myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, clinically significant transient ischemic attack, symptomatic pulmonary embolism, unexplained syncope, or long QT syndrome.
* Patient who is pregnant or breastfeeding.
* Patient with active bacterial, fungal, or viral infection, including but not limited to the use of antibiotics, antifungals, or antiviral agents at the time of Screening;
* Underlying medical conditions, laboratory abnormality, or alcohol or drug abuse or dependence that, in the Investigator's opinion, will be unfavorable for the administration of study treatment or affect the explanation of drug toxicity or adverse events; or insufficient compliance during the study according to Investigator's judgement; or
* Patient has experienced other severe acute or chronic medical or psychiatric conditions, including recent (within 1 year of signing informed consent/assent) or active suicidal ideation or behavior, or a laboratory abnormality that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the participant inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-10-13 (Estimated); Study Completion 2030-10-13 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of conducting a prospective single-center clinical trial of mirdametinib in patients with advanced NF1-mutant melanoma whose disease progresses during or after PD-1 antibody-based checkpoint inhibitor therapy. | 12 months
  This is a small pilot study to evaluate a feasibility of conducting a prospective single-center clinical trial of mirdametinib in patients with advanced NF1-mutant melanoma whose disease progresses during or after PD-1 antibody-based checkpoint inhibitor therapy. The primary endpoint is to enroll and treat 10 patients over a 12 month period. If there are at least 2 clinical responses among the 10 patients, the preliminary efficacy will be considered promising. Further discussions with the funding agency to expand the cohort to a total of 29 patients will then be planned.

SECONDARY OUTCOMES:
To evaluate the safety profile of mirdametinib in patients with advanced NF1-mutant melanoma | 2 years
  Descriptive statistics for safety will be presented using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. All on-study AEs, Grade 3-4 AEs, treatment-related AEs, Grade 3-4 treatment-related AEs, SAEs, AESIs, treatment-related SAEs, and AEs leading to dose reduction, dose interruption, and treatment discontinuation will be tabulated using worst grade per NCI CTCAE v 5.0 criteria by system organ class and preferred term. On-study lab and Grade 3-4 Lab Abnormalities will be summarized using baseline and worst grade NCI CTCAE v 5.0 criteria.
To evaluate preliminary clinical efficacy of mirdametinib in patients with advanced NF1-mutant melanoma whose disease has progressed while on or after previous immunotherapy | 12 months
  Descriptive statistics of enrollment rate, overall response rate, progression-free survival and overall survival will be performed. Endpoints for efficacy will include response rate by RECIST 1.1, progression-free survival, and survival by Kaplan-Meier analysis.
  If there are at least 2 clinical responses among the 10 patients, the preliminary efficacy will be considered promising.

CONTACTS AND LOCATIONS:
Locations (1):
- California Pacific Medical Center - Sutter Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon publication.